CLINICAL TRIAL: NCT02549924
Title: Effect of Administration of Resveratrol on Glycemic Variability in Individuals With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Brief Title: Effect of Administration of Resveratrol on Glycemic Variability in Individuals With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no financial support
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, Esperanza Martínez-Abundis, FACP, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERVGDM2
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Resveratrol; Glycemic Variability; MAGE
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Experimental): Individuals with T2DM inadequately controlled with metformin 2000 mg/day and A1C ≥7%.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Individuals with T2DM inadequately controlled with metformin 2000 mg/day and A1C ≥7%.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — Resveratrol capsules, 500 mg 3 times daily with the first bite of each meal
  Other Names: Trans-resveratrol
  Arms: Resveratrol
Drug: Placebo — Placebo capsules, 500 mg 3 times daily with the first bite of each meal
  Other Names: Calcined Magnesia
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus [ T2DM ] has quickly become the epidemic of the XXI century and challenging global health . Estimates of the World Health Organization [ WHO ] indicate that globally , from 1995 to date has nearly tripled the number of people living with diabetes mellitus [DM ]. Resveratrol has been extensively studied as a regulator of glucose through its antioxidant effects and protecting pancreatic β cells by activation of sirtuin -1 [ SIRT1 ] dependent deacetylase nicotinamide adenine diphosphate [ NAD ]. Therefore, it is important to know the effect of resveratrol on the glycemic variability [GV ] in patients with T2DM who are not in control with metformin monotherapy based.

DETAILED DESCRIPTION:
The objective is to evaluate the effect of administration of resveratrol on GV in individuals with T2DM inadequately controlled on metformin, for which we will conduct a double-blind trial, randomized, placebo control group, each group 11 male and female patients 30-60 years of age with T2DM inadequately controlled with metformin [2000 mg / day and glycosylated hemoglobin A1c (A1C) ≥% 7], with body mass index [BMI] form 25.0 to 34.9 kg / m2. Randomization will determine who will receive the intervention during the 8-week trial [resveratrol capsules, 500 mg 3 times daily with the first bite of each meal or approved placebo capsules], both groups also continue with metformin. The clinical findings and laboratory tests include a metabolic profile and biosafety, which will be made at baseline and at 8 weeks. Body weight, body fat, BMI and blood pressure will be determined during the initial and final visit, likewise, plasma glucose concentrations every hour recorded over 72 hours by continuous monitoring system outpatient glucose [MACG] via iPro ™ 2 [Medtronic MiniMed, Northridge] system, through which the mean amplitude of glucose excursions [MAGE] is calculated and AUC glucose, which will serve to assess the GV. Adverse events and adherence to treatment will be documented. Statistical analysis: Mann-Whitney U test, Wilcoxon and Fisher exact test. It is considered with significance at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* BMI from 25.0-34.9 kg/m2
* Diagnosis of T2DM
* Fasting plasma glucose >130 and <250 mg/dl at the time of scrutiny
* A1C between 7 and 10%
* Metformin monotherapy
* Written informed consent

Exclusion Criteria:

* Women pregnant or breastfeeding
* Untreated thyroid disease and/or uncontrolled hypertension [≥150 systolic and diastolic ≥90]
* Consumption of oral agents or other medications or supplements, unlike metformin, with proven properties that modify the behavior of glucose
* Total cholesterol >400 mg/dL
* Triglycerides ≥400 mg/dL
* Liver enzymes [ALT and AST] more than twice the normal range
* Glomerular filtration rate <60 mL/min [Cockcroft-Gault]

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve | 56 days
  Before and after intervention with ambulatory continuous glucose monitoring during 72 h, oxidase glucose iPro ™ 2
Mean amplitude of glucose excursions (MAGE) | 56 days
  Before and after intervention with ambulatory continuous glucose monitoring during 72 h, oxidase glucose iPro ™ 2

SECONDARY OUTCOMES:
Fasting plasma glucose | 56 days
  Before and after intervention by spectrophotometry
Postprandial glucose | 56 days
  Before and after intervention with ambulatory continuous glucose monitoring during 72 h, oxidase glucose iPro ™ 2
A1C | 56 days
  Before and after intervention by high-performance liquid chromatography
Total cholesterol | 56 days
  Before and after intervention by spectrophotometry
Triglycerides | 56 days
  Before and after intervention by spectrophotometry
High-density lipoprotein cholesterol | 56 days
  Before and after intervention by spectrophotometry
Low-density lipoprotein cholesterol | 56 days
  Friedewald formula
Very-low density lipoprotein | 56 days
  Friedewald formula
Alanine aminotransferase | 56 days
  Before and after intervention by spectrophotometry
Aspartate aminotransferase | 56 days
  Before and after intervention by spectrophotometry
Creatinine | 56 days
  Before and after intervention by spectrophotometry
Blood pressure | 56 days
  Before and after intervention using a digital manometer
Body and visceral fat % | 56 days
  Before and after intervention using a impedance bascule, Tanita MR

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez-Abundis, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico